CLINICAL TRIAL: NCT01695213
Title: A Randomized Comparative Study to Evaluate the Performance and Confirm the Safety of the Diocom Hip Syhstem in Cementless Hip Arthroplasty
Brief Title: RCT Comparing the DEXA Results of the HA-Omnifit Versus the Symax Uncemented Hip Stem
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Symax DEXA study; MEC 02-072 (Other: METC MUMC Maastricht)
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Patients With Osteoarthritis of the Hip Joint Elligable for a Uncemented Hipprosthesis
Keywords: uncemented hip; bone remodeling; DEXA; clinical evaluation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- HA-Omnifit (Active Comparator): Patients who receive a HA-Omnifit uncemented hip stem
  Interventions: Procedure: uncemented total hip arthroplasty
- Symax hip stem (Active Comparator): Patients with the Symax uncemented hip stem
  Interventions: Procedure: uncemented total hip arthroplasty

INTERVENTIONS:
Procedure: uncemented total hip arthroplasty

SUMMARY:
Thr purpose of this study is to compare the clinical and radiological results, as well as the femur bone density measurements of two uncemented total hip prostheses during 5 years of follow up.

DETAILED DESCRIPTION:
It is of great importance for the function of uncemented total hip arthroplasty that the anchorage of the prosthesis in the bone of the femur is sufficient. This is of great importance in the prevention of stress shielding of the bone and to insure tranfer of forces from the prosthesis to the femur.

The symax hip stem is developed to optimize stress tranfer to bone and insure mechanical stability.

In this study the symax hip stem is compared to the HA_Omnifit hip stem (a frequently used and long term evaluated uncemented hip prosthesis) During the fist two years of follow up DEXA mesurments of bone mineral density are performed. Also patient satisfaction, patient fuction score and radiological evaluation measurements are done during 5 years of follow up.

Our primary objective is: comparison of the short term bone remodelling surrounding the Symax hip stem to the short term remodeling surrounding the Stryker Omnifit HA hip stem measured by bone densitometry, clinical and radiographic evaluation.

ELIGIBILITY:
Inclusion Criteria:Male or non pregnant female patients >18 years

* Patient with degenerative or traumatic changes to hip requiring hip replacement
* Patient with BMI<35
* Patient signed informed consent

Exclusion Criteria:

* chronic anti-inflammatory medication use> 3 months
* revision surgery to the affected femur
* Cancer therapy including immunosuppression, chemotherapy and radiation
* Pathological fractures, delayed ossification or non-union is likely to occur

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
short term bone remodeling | 6 times within 2 years
  Bone remodeling is determined by measuring the Bone mineral density during time
complications and reoperations | during 5 years
  Reporting all complications and reoperations of the two different hip prostheses

SECONDARY OUTCOMES:
clinical performance | 9 times within 5 years
  Comparison of the clinical performance of the two different hip prostheses
Radiological evaluation | 9 times within 5 years
  Evaluation of Xrays according to the engh classifications

OTHER OUTCOMES:
patient satisfaction | 9 times within 5 years
  comparison of patient satisfaction between the two different prostheses

CONTACTS AND LOCATIONS:
Overall Officials: Lodewijk van Rhijn, Study Director — azM

REFERENCES:
- [Derived] ten Broeke RH, Tarala M, Arts JJ, Janssen DW, Verdonschot N, Geesink RG. Improving peri-prosthetic bone adaptation around cementless hip stems: a clinical and finite element study. Med Eng Phys. 2014 Mar;36(3):345-53. doi: 10.1016/j.medengphy.2013.12.006. Epub 2013 Dec 27. PMID 24378381